CLINICAL TRIAL: NCT06561256
Title: Effectiveness and Safety of Combination Therapy With Corticosteroids and JAK Inhibitors in Bullous Pemphigoid
Brief Title: JAK Inhibitors' Efficacy in Bullous Pemphigoid
Status: Completed | Type: Observational
Sponsor: Chao Ji (Other)
Responsible Party: Sponsor-Investigator, Chao Ji, Clinical Professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: FirstAHFujian123
Record Dates: First submitted 2024-08-15; First posted 2024-08-20 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Bullous Pemphigoid; Janus Kinase Inhibitor; Corticosteroids
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Janus Kinase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Janus Kinase Inhibitor — Janus Kinase Inhibitor in combination with corticosteroids

SUMMARY:
Bullous pemphigoid (BP) is an autoimmune subepidermal blistering skin disease that predominantly affects the elderly population, with rare cases reported in children and adolescents. BP is characterized by circulating antibodies that target the hemidesmosomal proteins bullous pemphigoid Antigen 1 (BPAg1 or BP230) and bullous pemphigoid Antigen 2 (BPAg2 or BP180/collagen XVII) located at the dermal-epidermal junction. The first-line treatment of BP includes topical or systemic use of corticosteroids. For refractory cases or when corticosteroids are contraindicated or to minimize adverse effects, adjunct therapies such as immunosuppressants (e.g. azathioprine, cyclosporine), dapsone, tetracycline antibiotics combined with niacinamide, intravenous immunoglobulins (IVIG), and plasma exchange are employed. Recent research has explored the use of biologic agents to treat refractory BP, including anti-CD20 monoclonal antibodies, anti-IgE monoclonal antibodies, and anti-interleukin monoclonal antibodies, showing promising outcomes. Nevertheless, effectively managing BP remains a challenge.

The Janus kinase (JAK)-signal transducer and activator of transcription (STAT) pathway has been implicated as a key driver in many inflammatory diseases. Recently, a class of drugs targeting this pathway, known as JAK inhibitors, has been developed. Some studies have investigated the efficacy and safety of JAK inhibitors combination with corticosteroids in BP treatment. In this retrospective study, the investigators conducted a comparative analysis to evaluate the efficacy and safety of JAK inhibitors combination With corticosteroids for patients diagnosed with moderate-to-severe bullous pemphigoid.

DETAILED DESCRIPTION:
This study will conduct a retrospective review of patients with Bullous pemphigoid in the Department of Dermatology of the First Affiliated Hospital of Fujian Medical University. Researchers will initially screen patients based on the inclusion and exclusion criteria through their respective hospital's medical record systems at the beginning of the study. All enrolled patients will be followed for a duration of 48 weeks. This study will include approximately 300 patients with moderate to severe BP.

The Primary outcomes were the time to cease of new lesions, time to achieve minimal therapy, the cumulative amount of corticosteroids (at the time of achieving minimal therapy). The Secondary outcomes were the scores of BPDAI (week 0, week 2, and week 4). the scores of itching Numeric Rating Scale (NRS) (week 0, week 2, and week 4). the level of IgE (week 0, week 2) and eosinophil percentage (Eos%) (week 0, week 2). the clinical remissions at week 24 and week 48. Adverse events: all treatment-related adverse events (AEs) were assessed.

The statistical analysis was performed using GraphPad Prism software 10.0 and SPSS 29.0. Categorical variables were presented as frequencies and percentages. Continuous variables were represented as means and standard deviations (SD) or as medians and interquartile ranges (IQR). Absolute and relative frequencies were used to describe qualitative variables. Groups were compared using chi-square test for qualitative variables and independent sample t-test or analysis of variance (ANOVA) for quantitative variables with symmetric distribution. The Mann-Whitney U test or Kruskal-Wallis test were used for quantitative variables with skewed distributions. P< 0.05 was considered statistically significant.

Upon completion, the study will analyze the collected data and to assess the efficacy and safety of the combination of Janus kinase inhibitors and corticosteroids in treatment of BP.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Bullous pemphigoid;
2. Moderate to severe bullous pemphigoid； The disease severity was measured using the Bullous Pemphigoid Disease Area Index (BPDAI) score and was classified into mild (BPDAI ≤ 19), moderate (20 ≤ BPDAI ≤ 56), and severe (BPDAI ≥ 57).
3. Moderate to severe BP received JAK Inhibitors combination with corticosteroids therapy；

Exclusion Criteria:

1. Patients diagnosed with malignant neoplasms
2. Previous administration with biologics within 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All enrolled patients will be followed for a duration of 48 weeks. This study will include approximately 300 patients with moderate to severe BP. The Primary outcomes were the time to cease of new lesions, time to achieve minimal therapy, the cumulative amount of corticosteroids (at the time of achieving minimal therapy). The Secondary outcomes were the scores of BPDAI (week 0, week 2, and week 4). the scores of itching Numeric Rating Scale (NRS) (week 0, week 2, and week 4). the level of IgE (week 0, week 2) and eosinophil percentage (Eos%) (week 0, week 2). the clinical remissions at week 24 and week 48. Adverse events: all treatment-related adverse events (AEs) were assessed.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Time to cease of new lesions | 2022.01.01-2024.07.31
  The time from baseline to cease of new blister formation.
Time to achieve minimal therapy. | 2022.01.01-2024.07.31
  Minimal therapy defined as ≤ 0.1 mg/kg/d of prednisone (or equivalent) or 20 g/wk of clobetasol propionate and/or minimal adjuvant or maintenance therapy
The cumulative amount of methylprednisolone (at the time of achieving minimal therapy). | 2022.01.01-2024.07.31
  The cumulative amount of methylprednisolone from baseline to the time of achieving minimal therapy

SECONDARY OUTCOMES:
The scores of BPDAI | 2022.01.01-2024.07.31
  the Bullous Pemphigoid Disease Area Index (BPDAI) scores and was classified into mild (BPDAI ≤ 19), moderate (20 ≤ BPDAI ≤ 56), and severe (BPDAI ≥ 57). This study included patients with moderate to severe BP.
The scores of itching Numeric Rating Scale (NRS) | 2022.01.01-2024.07.31
  The patient is asked to rate their current level of itching on this 0-10 scale. 0 - No itching 1-3 - Mild itching 4-6 - Moderate itching 7-10 - Severe itching. This NRS score for itching can help healthcare providers assess the severity of the patient's itching, track changes over time, and guide appropriate treatment interventions.
Adverse events | 2022.01.01-2024.07.31
  All treatment-related adverse events (AEs) were assessed.
Clinical remissions | 2022.01.01-2024.07.31
  Partial remission on minimal therapy: presence of transient new lesions that heal within 1 week while patient is receiving minimal therapy for at least 2 months Complete remission on minimal therapy: absence of new or established lesions or pruritus while patient is receiving minimal therapy for at least 2 months Partial remission off therapy: presence of transient new lesions that heal within 1 week without treatment while patient is off all BP therapy for at least 2 months.
  Complete remission off therapy: absence of new or established lesions or pruritus while patient is off all BP therapy for at least 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Ji, PhD, Study Chair — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fujian, Fuzhou, China

IPD SHARING:
Plan to Share IPD: No